CLINICAL TRIAL: NCT02430831
Title: Randomized Controlled Trial Testing the Effect of Milk Formula Supplemented With L. Reuteri on Crying Time in Colicky Infants Less Than 3 Months Old
Brief Title: Effect of Milk Formula Supplemented With L. Reuteri on Crying Time in Colicky Infants Less Than 3 Months Old
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bari (Other)
Collaborators: Antonio Di Mauro (Unknown); Ruggiero Francavilla (Unknown); Lorenzo Trovè (Unknown)
Responsible Party: Principal Investigator, Flavia Indrio, MD, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VF/FC
Record Dates: First submitted 2015-03-31; First posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Infantile Colic
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reuteri group (Active Comparator): Milk formula added with probiotic L reuterii DSM 17938
  Interventions: Dietary Supplement: Nidina
- Placebo (Placebo Comparator): Milk formula without probiotic L reuterii DSM 17938
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nidina
  Arms: Reuteri group
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Study type:

Randomized controlled trial with two parallel arms Objectives

Primary : Demonstrate that daily supplementation of colicky infants with Nidina formula containing L. reuteri DSM 17938 decreases the daily crying duration at 21 days Secondary : Evaluate the effects of daily supplementation of colicky infants with Nidina formula containing L. reuteri DSM 17938 measured as

1. the number of "responders" or the "treatment success" (ie infants for which defined as the percentage of children achieving a reduction in the daily average crying time >50% in 3 weeks. (day 1 to day 21 of the study)
2. maternal depression and family functioning scoring

DETAILED DESCRIPTION:
Inclusion criteria :

* less then 12 weeks of age
* term infant (≥ 38 weeks gestational age)
* birth weight > 2,500g
* infantile colic diagnosed according to modified Wessel's criteria, i.e. crying more than an average of 180 min/day during the 3 days prior to enrollment.
* parental motivation to postpone changes in the infant feeding mode, unless necessary

Exclusion criteria:

* birth weight less than 2500 g
* failure to thrive
* chronic illness or major medical problem
* gastrointestinal disease
* cow's milk allergy ( confirmed prior to exclusion; difficult to diagnose so early ??)
* use of any antibiotic or probiotic in the week (7 days) prior to enrollment
* use of proton pump inhibitors in the week (7 days) prior to enrollment
* if breastfeeding, use of probiotic by the mother in the week (7 days) prior to enrollment
* infant receiving solid foods (such as cereals, mashed fruits or vegetable purée)
* change of feeding mode planned by parents during the study period

Randomization and blinding: to be written by the CRO, according to its own procedures.

Extreme caution should be given to blinding. Methods should give full certainty that blinding was perfect at the subject (parent) level, but also at the pediatrician and with all involved personnel.

Randomization should be done according to 3 feeding modes :

* "breast feeding: only breast, except for 2 bottle feedings a week,
* "formula fed": only formula except two breast feeding a week,
* "mixed feeding": all the remaining

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria :
* less then 12 weeks of age
* term infant (≥ 38 weeks gestational age)
* birth weight > 2,500g
* infantile colic diagnosed according to modified Wessel's criteria, i.e. crying more than an average of 180 min/day during the 3 days prior to enrollment.
* parental motivation to postpone changes in the infant feeding mode, unles

Exclusion Criteria:

* - birth weight less than 2500 g
* failure to thrive
* chronic illness or major medical problem
* gastrointestinal disease
* cow's milk allergy ( confirmed prior to exclusion; difficult to diagnose so early ??)
* use of any antibiotic or probiotic in the week (7 days) prior to enrollment
* use of proton pump inhibitors in the week (7 days) prior to enrollment
* if breastfeeding, use of probiotic by the mother in the week (7 days) prior to enrollment
* infant receiving solid foods (such as cereals, mashed fruits or vegetable purée)
* change of feeding mode planned by parents during the study period

Max Age: 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Daily Crying duration | three days
  The average crying time in minutes per day measured on day 19, 20, and 21 between active and placebo groups.

SECONDARY OUTCOMES:
Rate of success (decrease in mean daily crying time) | 3 days
  Percentage of infants in the active group compared to the placebo group in whom the mean of daily crying time of the days 19, 20 and 21 decreased by 50% compared to the three days prior to recruitment.
Family functional score (family functioning scale) | one day
  The score achieved in the family functioning scale at day 21.
Mother depression (mother depression Scale) | One day
  The score achieved in the mother depression Scale at day 21.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Indrio, MD, Principal Investigator — University of Bari
Locations (1):
- University of Bari, Bari, BA, Italy